CLINICAL TRIAL: NCT03543943
Title: Achilles Tendon Elongation and Gait Pattern After Rupture: A Three Armed Randomized Controlled Trial Comparing an Individualized Treatment Algorithm vs. Operative or Non-operative Treatment.
Brief Title: Achilles Tendon Elongation and Gait Pattern After Rupture.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Maria Swennergren Hansen, Principal Investigator, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Achilles HVH RCT
Record Dates: First submitted 2018-05-03; First posted 2018-06-01 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Achilles Tendon Rupture

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The posterior site of the achilles tendon region is covered by dark tape during the functional assesments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Individualized treatment (Experimental): The ruptured achilles tendon is examined by ultrasonography. If the overlap of the tendon ends is less than 25 % or the tendon is elongated 7 % or more the patient receives conventional open operative treatment. The tendon is sutured with double fiberwire size 2 a.m. Kessler under prophylactic Dicloxacillin 2 g and in local anesthesia or alternatively popliteal or spinal block. The injured leg is placed in a circulated below the knee cast after surgery. The ankle is held at maximal plantar flexion. Weight bearing is not allowed. After 3 weeks the cast is removed and the injured leg is transferred to a functional brace with 3 heel wedges. The patient will follow standard functional rehabilitation and the follow-up evaluations.
  Interventions: Procedure: Individualized treatment of Acute Achilles tendon rupture.
- Control group 1 (Active Comparator): For the patients allocated to non-operative treatment the injured leg is placed in a circulated below the knee cast from the time of the first appointment in the Outpatients Department. The ankle is held at maximal, unforced plantar flexion. Weight bearing is not allowed and the patient should walk with the aid of crutches. After 3 weeks from initiated treatment in the Emergency Department the cast is removed in the Outpatients Department and the injured leg is transferred to a functional brace (Walker boot) with 3 heel wedges promoting 20 degrees plantar flexion over the ankle. The patient will follow standard functional rehabilitation and the follow-up evaluations.
  Interventions: Procedure: Non-operative treatment
- Control group 2 (Active Comparator): The tendon is sutured with double fiberwire size 2 a.m. Kessler under prophylactic Dicloxacillin 2 g and in local anesthesia or alternatively popliteal or spinal block. The injured leg is placed in a circulated below the knee cast from the time of the first appointment in the Outpatients Department. The ankle is held at maximal, unforced plantar flexion. Weight bearing is not allowed and the patient should walk with the aid of crutches. After 3 weeks from initiated treatment in the Emergency Department the cast is removed in the Outpatients Department and the injured leg is transferred to a functional brace (Walker boot) with 3 heel wedges promoting 20 degrees plantar flexion over the ankle. The patient will follow standard functional rehabilitation and the follow-up evaluations.
  Interventions: Procedure: Operative treatment

INTERVENTIONS:
Procedure: Individualized treatment of Acute Achilles tendon rupture. — The most proximal border of the calcaneus and the most distal point of the musculotendinous junction of the medial gastrocnemius muscle is identified and marked on the skin. These two points on the un-injured leg defines the original length of the total Achilles tendon [1]. The difference in length between the injure and the un-injured leg determines elongation for the ruptured Achilles tendon. The relative elongation of the ruptured tendon together with overlap of the tendon ends on the cross-sectional area determines the treatment for the patients receiving individualized treatment: 1) patients with 0-6% elongation of the tendon and a minimum of 25% tendon are treated non-operatively 2) patients with 7% elongation or more or less than 25% tendon overlap are treated operatively.
  Arms: Individualized treatment
Procedure: Non-operative treatment — Circulated cast below the knee in maximal, unforced plantar flexion over the ankel.
  Arms: Control group 1
Procedure: Operative treatment — Open surgery with suture of the ruptured achilles tendon prior to circulated cast below the knee in maximal, unforced plantar flexion over the ankel.
  Arms: Control group 2

SUMMARY:
The objective of this study is to determine if Achilles tendon elongation and gait pattern differ between patients treated using an individualized treatment algorithm and patients treated as usual (two control groups; patients treated operatively and non-operatively).

The individualized treatment algorithm is based on ultrasonographic status of tendon overlap and Copenhagen Achilles Length Measure (1). Patients are allocated for operative treatment if there the tendon overlap is less than 25 % or the tendon is elongated with 7% or more compared to the healthy, contralateral achilles tendon.

ELIGIBILITY:
Inclusion Criteria:

* Appointment in the Outpatients Department within 4 days of injury.
* Total Achilles tendon rupture.
* Initial treatment with split cast with the ankle in maximal plantar flexion must be started within 24 hours of injury.
* The patient must be expected to be able to attend rehabilitation and postexamination.
* The patient must be able to speak and understand Danish.
* The patient must be able to give informed consent.

Exclusion Criteria:

* Rupture of the Achilles tendon either at the insertion on the calcaneus or at musculotendinous junction of the triceps surae.
* Previous rupture of the Achilles tendon in any of the two legs.
* Treated with fluoroquinolones or corticosteroids within the last 6 months.
* In medical treatment of diabetes.
* Suffers from rheumatic disease.
* Other conditions prior to the injury resulting in reduced function of any of the two legs.
* Contra-indication for surgery: severe arthrosclerosis with no palpable pulse in the foot, broken skin in the Achilles region of the injured leg.
* Inability to lie in prone position on the operating table.
* Terminal illness or severe medical illness: American Society of Anaesthesiologists physical status classification score higher than or equal to 3.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Three-Dimensional Gait Analysis: Ankle peak power during push-off. | 12 months after started treatment.
  Reflective markers placed on the patients skin with tape on specific anatomical locations, in total 19 markers. The reflective markers are being filmed by 8 infrared cameras hanging on the walls around the laboratory. Thereby, the joint angles during gait will be measured, and, in combination with the ground reaction forces from two force plates embedded in the floor, the joint moments and powers will be calculated.

SECONDARY OUTCOMES:
Copenhagen Achilles Length Measure | 6 and 12 months after started treatment.
  The examination of both the total and the free part of the achilles tendon of both the injured and un-injured leg is performed. The total length of the tendon is defined under the description of the intervention. The free part of the achilles tendon is defined as the distance between the proximal border of calcaneus and the musculotendinous junction of the soleus muscle and the achilles tendon. The method will be used both diagnostically for the individualized treatment and as a secondary endpoint.
Three-Dimensional Gait Analysis: Ankle peak power during push-off | 6 months after started treatment.
  Reflective markers placed on the patients skin with tape on specific anatomical locations, in total 19 markers. The reflective markers are being filmed by 8 infrared cameras hanging on the walls around the laboratory. Thereby, the joint angles during gait will be measured, and, in combination with the ground reaction forces from two force plates embedded in the floor, the joint moments and powers will be calculated.
Three-Dimensional Gait Analysis: Maximal dorsiflexion in the stance phase. | 6 and 12 months after started treatment.
  Reflective markers placed on the patients skin with tape on specific anatomical locations, in total 19 markers. The reflective markers are being filmed by 8 infrared cameras hanging on the walls around the laboratory. Thereby, the joint angles during gait will be measured, and, in combination with the ground reaction forces from two force plates embedded in the floor, the joint moments and powers will be calculated.
Three-Dimensional Gait Analysis: stiffness of the plantar flexor musculo-tendinous complex during dorsiflexion. | 6 and 12 months after started treatment.
  Reflective markers placed on the patients skin with tape on specific anatomical locations, in total 19 markers. The reflective markers are being filmed by 8 infrared cameras hanging on the walls around the laboratory. Thereby, the joint angles during gait will be measured, and, in combination with the ground reaction forces from two force plates embedded in the floor, the joint moments and powers will be calculated.
Three-Dimensional Gait Analysis: time of heel-lift | 6 and 12 months after started treatment.
  Reflective markers placed on the patients skin with tape on specific anatomical locations, in total 19 markers. The reflective markers are being filmed by 8 infrared cameras hanging on the walls around the laboratory. Thereby, the joint angles during gait will be measured, and, in combination with the ground reaction forces from two force plates embedded in the floor, the joint moments and powers will be calculated.
Three-Dimensional Gait Analysis: jumping up and down | 6 and 12 months after started treatment.
  Reflective markers placed on the patients skin with tape on specific anatomical locations, in total 19 markers. The reflective markers are being filmed by 8 infrared cameras hanging on the walls around the laboratory. Thereby, the joint angles during gait will be measured, and, in combination with the ground reaction forces from two force plates embedded in the floor, the joint moments and powers will be calculated.
Balance measurement | 6 and 12 months after started treatment.
  The postural sway with patient standing on a force plate in the gait laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Maria S Hansen, PT, MSc, Principal Investigator — Copenhagen University Hospital, Amager-Hvidovre
Locations (1):
- Department of Physiotherapy and Orthopedical surgery, Copenhagen University Hospital, Amager-Hvidovre, Copenhagen, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No
There is no plan of sharing data with researchers not already included in this study.

REFERENCES:
- [Background] Barfod KW, Riecke AF, Boesen A, Hansen P, Maier JF, Dossing S, Troelsen A. Validation of a novel ultrasound measurement of achilles tendon length. Knee Surg Sports Traumatol Arthrosc. 2015 Nov;23(11):3398-406. doi: 10.1007/s00167-014-3175-2. Epub 2014 Jul 20. PMID 25038882